CLINICAL TRIAL: NCT01754545
Title: Prophylactic Plasma Infusion Therapy for Congenital Thrombotic Thrombocytopenic Purpura
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: altered situation in study population; not enough patients meeting enrollment criteria
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 133995
Record Dates: First submitted 2012-12-12; First posted 2012-12-21 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-12

CONDITIONS: Purpura, Thrombotic Thrombocytopenic
Keywords: Infusions, Intravenous; Plasma; ADAMTS-13 protein, human
MeSH Terms: conditions — Purpura, Thrombotic Thrombocytopenic | interventions — Solvents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Octaplas infusion and placebo (group 1) (Experimental): Active treatment with randomly assigned 400 ml octaplas intravenously 2-3 times a week and 400 ml placebo (for octaplas)intravenously 2-3 times a week over two weeks.
  Interventions: Drug: Octaplas infusion and placebo (group 1)
- Octaplas infusion and placebo (group 2) (Experimental): Active treatment with randomly assigned 400 ml octaplas intravenously once and 400 ml placebo (for octaplas)intravenously twice in two separate intervention weeks
  Interventions: Drug: Octaplas infusion and placebo (group 2)

INTERVENTIONS:
Drug: Octaplas infusion and placebo (group 1) — Intervention period is Monday-Friday in two following weeks. Active treatment with Octaplas is given 2-3 times each week and placebo is given the other 2-3 days of intervention each week. Route of administration is intravenously.
  Other Names: ATC B05A A02; Solvent/detergent plasma; Human plasma
  Arms: Octaplas infusion and placebo (group 1)
Drug: Octaplas infusion and placebo (group 2) — Intervention period is Monday-Wednesday in two separate weeks (minimum of three weeks between intervention weeks). Active treatment with Octaplas is given once and placebo is given twice each week. Route of administration is intravenously.
  Other Names: ATC B05A A02; Solvent/detergent plasma; Human plasma
  Arms: Octaplas infusion and placebo (group 2)

SUMMARY:
Congenital thrombotic thrombocytopenic purpura (TTP), also called Upshaw-Schulman Syndrome or hereditary or familial TTP is a rare, but severe disease. The purpose of this study is to determine how infusions of plasma to patients with congenital TTP correlate with symptoms and signs of activity of the disease, and to determine why some patients need more frequent infusions of plasma than others to prevent acute attacks of the disease.

DETAILED DESCRIPTION:
Patients with congenital TTP have an inherited lack of function or amount of a protein in plasma called ADAMTS13, that otherwise is responsible for cleaving large von Willebrand-molecules into smaller parts. The patients suffer recurrent attacks of clotting of small blood vessels, that can cause damage to major organs, including the central nervous system. Acute attacks can be treated successfully with infusions of human plasma, and some patients also receive regular plasma therapy for prevention of acute attacks. A small group of patients receive preventive plasma infusions twice or more weekly, indicating a much higher need for plasma than what is otherwise recommended for preventive therapy. Do these patients have an ongoing activity of their disease despite a stimulus? Or a higher turn-over of transfused ADAMTS13? Have these patients developed antibodies against transfused ADAMTS13? Are any symptoms correlated with signs of disease activity?

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of congenital TTP
* On regular prophylactic plasma treatment: > Once weekly (group 1) or >1 <3 times monthly (group 2)
* Between 18 and 65 years
* Capable of understanding and complying with the protocol

Exclusion Criteria:

* Pregnancy
* Acute bout of TTP requiring daily plasma infusions or -exchange for more than 3 days, within the last 2 weeks before intervention period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
A composite score of clinical and biochemical signs of disease activity | 4 hours and 24 hours after intervention
  Biochemical signs of disease activity are scored by measurements of lactate dehydrogenase, hemoglobin, platelet counts and ADAMTS13 activity.
  Clinical signs of disease activity are measured by an evaluator's score and subjects symptom screening

SECONDARY OUTCOMES:
ADAMTS13 activity half-life | 4 hours and 24 hours after intervention
  Calculation of half-life of ADAMTS13 activity based on serial measurements of ADAMTS13 activity before and after plasma infusions
ADAMTS13 allo-antibodies | At baseline
  Presence of allo-antibodies towards ADAMTS13

CONTACTS AND LOCATIONS:
Overall Officials: Anne S von Krogh, MD, Principal Investigator — St. Olavs Hospital